CLINICAL TRIAL: NCT00310531
Title: A Multicenter, Double-Blind, Double-Dummy, Randomized, Active- Controlled, 3-Year Study to Evaluate the Antiresorptive Efficacy, Safety and Tolerability of a Ultra-Low Dose Estradiol Transdermal Delivery System Releasing 0.014 mg / Day Versus Oral Raloxifene Hydrochloride 60 mg / Day - as a Therapy for the Prevention of Osteoporosis in Postmenopausal Female Osteopenic Patients.
Brief Title: 3-year Study of Menostar Versus Evista to Prevent Osteoporosis in Post-menopausal Women
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 91213; 306871
Record Dates: First submitted 2006-03-31; First posted 2006-04-04 (Estimated); Last update posted 2014-12-30 (Estimated); Status verified 2014-12

CONDITIONS: Osteopenia
MeSH Terms: conditions — Bone Diseases, Metabolic | interventions — Estradiol; Raloxifene Hydrochloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1 (Experimental)
  Interventions: Drug: Menostar (Estradiol, BAY86-5435)
- Arm 2 (Active Comparator)
  Interventions: Drug: Raloxifene

INTERVENTIONS:
Drug: Menostar (Estradiol, BAY86-5435) — Menostar (estradiol transdermal delivery system (SHP00577E), 0.014 mg/day)
  Arms: Arm 1
Drug: Raloxifene — Raloxifene tbl. (60 mg/day)
  Arms: Arm 2

SUMMARY:
The aim of this trial is to investigate whether the Menostar patch is as safe and effective in the prevention of bone loss in postmenopausal women as raloxifen, a drug already registered for prevention and treatment of osteoporosis.

DETAILED DESCRIPTION:
The study has previously been posted by Schering AG, Germany. Schering AG, Germany has been renamed to Bayer Schering Pharma AG, Germany.Bayer Schering Pharma AG, Germany is the sponsor of the trial.

ELIGIBILITY:
Inclusion Criteria:

* Last (regular) menstrual period more than 5 years ago
* Relative good state of health
* Intact, normal uterus

Exclusion Criteria:

* Bone and musculoskeletal diseases
* Clinically significant vertebral fracture within the last 12 months
* Pre-existing cardiovascular disease (e.g. uncontrolled high/low blood pressure, stroke, thromboembolic event etc)
* Uncontrolled diabetes mellitus (or treated with insulin)
* Uncontrolled thyroid disorders
* Relevant renal disorder or significant liver dysfunction (including cholestasis)
* History of alcohol or drug abuse
* History of immobilization of more than 2 months in the last 6 months
* Smoking of more than 10 cigarettes per day
* Unexplained uterine bleeding
* Known or suspected malignant or premalignant disease (e.g. cancer of breast or uterus, melanoma)

Ages: 55 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Actual)
Dates: Start 2004-02; Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
Percentage change in Bone Mineral Density at the lumbar spine | after 3 years

SECONDARY OUTCOMES:
Percentage change in Bone Mineral Density of the hip | after 3 years
Percentage change in biochemical markers of bone turnover | after 6 months
Proportion of patients with hot flushes | after 3 year
Change in Women's Health Questionnaire | after 2 years
Proportion of patients with an abnormal endometrial biopsy | after 3 years
Pharmacogenetic analysis | after 2 years
Digital breast density analysis | after 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer